CLINICAL TRIAL: NCT06645392
Title: COMPARATIVE STUDY BETWEEN TERNAMIAN BLADELESS TROCAR ENTRY and VISUAL TRANSPARENT BLADED TROCAR ENTRY in LAPAROSCOPIC PROCEDURES; a PROSPECTIVE RANDOMIZED CONTROLLED TRIAL
Brief Title: COMPARATIVE STUDY BETWEEN TERNAMIAN BLADELESS TROCAR ENTRY and VISUAL TRANSPARENT BLADED TROCAR ENTRY in LAPAROSCOPIC PROCEDURES
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abdalla, Dr. Marwa Abdalla, Cairo University
Other Study IDs: LAPAROSCOPIC TROCARS
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Laparoscopic Entry Technique
Keywords: Visual - Transparent - Bladed-Bladeless - Ternamian - trocar laparoscopy).

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A, (Visual transparent bladed trocar group): visual transparent bladed trocar of diameter 10 mm is used for abdominal entry; the assistant holds the laparoscope mounted in the cannula of the trocar, and the surgeon lowers the unit (laparoscope and mounted cannula) deep into the umbilical wound where the surgeon uses the muscles of the dominant wrist to rotate the cannula clockwise while keeping the forearm horizontal the patient's abdomen. Downwards axial pressure during rotation is kept to a minimum. Rotation serves to lift the anterior abdominal wall and transpose successive tissue layers onto the cannula's outer thread. The white anterior rectus fascia, red rectus fascia, pearly white posterior rectus fascia, yellowish preperitoneal space, and transparent greyish peritoneal membrane are all observed sequentially on the monitor. Further clockwise rotation parts the peritoneal membrane radially to advance the cannula incrementally into the peritoneal cavity under direct visual control while avoiding cannula overshot
  Interventions: Device: visual transparent bladed trocar of
- Group B ( Ternamian bladeless trocar group): Ternamian bladeless trocar of diameter 10 mm is used for abdominal entry; this trocar is hollow in which a laparoscope is loaded for the distal crystal tip to transmit real-time monitor images while transecting abdominal wall tissue layers. The assistant holds the laparoscope during entry allowing the wrist to move freely while the surgeon applies significant axial thrust through the dominant upper body muscles while twisting the handle to advance the trocar tip and dissect successive tissue layers on its way towards the abdomen. A considerable axial force is applied by the surgeon for the retention of the push-through trocar design with no mechanism to offset overshoot.
  Interventions: Device: Ternamian bladeless trocar

INTERVENTIONS:
Device: visual transparent bladed trocar of — visual transparent bladed trocar of diameter 10 mm and Ternamian bladeless trocar of diameter 10 mm
  Groups: Group A, (Visual transparent bladed trocar group)
Device: Ternamian bladeless trocar — Ternamian bladeless trocar of diameter 10 mm
  Groups: Group B ( Ternamian bladeless trocar group)

SUMMARY:
To compare the efficacy and safety between Ternamian bladeless trocar entry and visual, transparent bladed trocar entry in laparoscopic procedures. A prospective randomized controlled study will be conducted among 100 female patients who will be admitted to the department of Gynecology and Obstetrics at Kasr Alainy university hospital for diagnostic and/or therapeutic laparoscopic intervention. Patients will be randomly assigned (1:1) using computer-generated random numbers to undergo laproscopic entry either by the visual transparent bladed trocar or the Ternamian bladeless trocar.

Main outcome measures: entry time of trocar entry in seconds and visceral or major vascular injury during trocar entry.

DETAILED DESCRIPTION:
To compare the efficacy and safety between Ternamian bladeless trocar entry and visual transparent bladed trocar entry in laparoscopic procedures. A prospective randomized controlled study will be conducted among 100 female patients who were admitted to the department of Gynecology and Obstetrics at Kasr Alainy university hospital for diagnostic and/or therapeutic laparoscopic intervention. Patients were randomly assigned (1:1) using computer-generated random numbers to undergo laproscopic entry either by the visual transparent bladed trocar or the Ternamian bladeless trocar. Entry time in seconds starting from the moment the trocar is applied through the umbilical incision to the moment the peritoneal cavity is entered, guided by transmitted images on the monitor, will be used to assess the efficacy of the used trocar type. Complications including major vessel injury or visceral injury that maybe encountered during laparoscopic entry could be immediately detected in both groups through the transmitted in time monitor images to assess safety of the used trocar type.

Main outcome measures: entry time of trocar entry in seconds and visceral or major vascular injury during trocar entry.

ELIGIBILITY:
Inclusion Criteria:

* included patients aged from 20 to 50 years old with uterine and/or adnexal benign lesions, infertility, or chronic pelvic pain indicated for diagnostic and/or therapeutic intervention, and with a body mass index (BMI) less than 40.

Exclusion Criteria:

* included patients who have had a history suggestive of pelvic adhesions as previous 4 or more laparotomies, a history of bleeding tendency, and patients with suspected pelvic malignancies.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — inclusion criteria included patients aged from 20 to 50 years old with uterine and/or adnexal benign lesions, infertility, or chronic pelvic pain indicated for diagnostic and/or therapeutic intervention, and with a body mass index (BMI) less than 40.
Study Population: Female patients aged from 20 to 50 years old with uterine and/or adnexal benign lesions, infertility, or chronic pelvic pain indicated for diagnostic and/or therapeutic intervention, and with a body mass index (BMI) less than 40.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
laparoscopic entry time | 6 months
  Time of entry was accurately estimated in both groups in seconds starting from the moment the trocar is applied through the umbilical incision to the moment the peritoneal cavity is entered guided by transmitted images on the monitor.

SECONDARY OUTCOMES:
Entry complications | 6 months
  Complications including major vessel injury or visceral injury that may be encountered during laparoscopic entry could be immediately detected in both groups through the transmitted in time monitor images.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Teaching Hospital, Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Laparoscopic primary entry: visual transparent bladed trocar entry vs Ternamian bladeless trocar entry
Supporting Information: Study Protocol
Time Frame: from now forever
Access Criteria: everyone